CLINICAL TRIAL: NCT05116202
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Melanoma (Morpheus-Melanoma)
Brief Title: A Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Melanoma (Morpheus-Melanoma)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO43328
Record Dates: First submitted 2021-10-22; First posted 2021-11-10 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab; atezolizumab; Tiragolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Nivolumab + Ipilimumab (Active Comparator): Cohort 1 participants in the nivolumab plus ipilimumab arm will receive treatment for 2 cycles (6 weeks) on Day 1 of each cycle (cycle length 21 days) until surgery, or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Cohort 1: RO7247669 2100 mg (Experimental): Cohort 1 participants in the RO7247669 arm will receive treatment for 2 cycles (6 weeks) until surgery, or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: RO7247669 2100 mg
- Cohort 1: + Atezolizumab + Tiragolumab (Experimental): Cohort 1 participants in the atezolizumab plus tiragolumab arm will receive treatment for 2 cycles (6 weeks) until surgery, or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Cohort 1: RO7247669 2100 mg + Tiragolumab (Experimental): Cohort 1 participants in the RO7247669 plus tiragolumab arm will receive treatment for 2 cycles (6 weeks) until surgery, or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: RO7247669 2100 mg; Drug: Tiragolumab
- Cohort 2: RO7247669 2100 mg + Tiragolumab (Experimental): Cohort 2 participants in RO7247669 plus tiragolumab arm will receive treatment until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: RO7247669 2100 mg; Drug: Tiragolumab
- Cohort 1: RO7247669 600 mg (Experimental): Cohort 1 participants in the RO7247669 arm will receive treatment for 2 cycles (6 weeks) until surgery, or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: RO7247669 600 mg
- Cohort 1: RO7247669 600 mg + Tiragolumab (Experimental): Cohort 1 participants in the RO7247669 plus tiragolumab arm will receive treatment for 2 cycles (6 weeks) until surgery, or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: Tiragolumab; Drug: RO7247669 600 mg

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be administered at a dose of 3 mg/kg IV on Day 1 of each 21 day cycle.
  Arms: Cohort 1: Nivolumab + Ipilimumab
Drug: Ipilimumab — Ipilimumab will be administered at a dose of 1 mg/kg by IV on Day 1 of each 21 day cycle.
  Arms: Cohort 1: Nivolumab + Ipilimumab
Drug: RO7247669 2100 mg — RO7247669 will be administered at a dose of 2100 mg by IV infusion on Day 1 of each 21 day cycle.
  Arms: Cohort 1: RO7247669 2100 mg; Cohort 1: RO7247669 2100 mg + Tiragolumab; Cohort 2: RO7247669 2100 mg + Tiragolumab
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg IV on Day 1 of each 21 day cycle.
  Other Names: Tecentriq, RO5541267
  Arms: Cohort 1: + Atezolizumab + Tiragolumab
Drug: Tiragolumab — Tiragolumab will be administered at a dose of 600 mg IV on Day 1 of each 21 day cycle.
  Other Names: RO7092284
  Arms: Cohort 1: + Atezolizumab + Tiragolumab; Cohort 1: RO7247669 2100 mg + Tiragolumab; Cohort 1: RO7247669 600 mg + Tiragolumab; Cohort 2: RO7247669 2100 mg + Tiragolumab
Drug: RO7247669 600 mg — RO7247669 will be administered at a dose of 600 mg by IV infusion on Day 1 of each 21 day cycle.
  Arms: Cohort 1: RO7247669 600 mg; Cohort 1: RO7247669 600 mg + Tiragolumab

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of treatment combinations in cancer immunotherapy (CIT)-naive participants with resectable Stage III melanoma (Cohort 1) and in participants with Stage IV melanoma (Cohort 2). The study is designed with the flexibility to open new treatment arms as new treatments become available, close existing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, and modify the participant population.

ELIGIBILITY:
Inclusion Criteria for Cohort 1:

* ECOG performance status (PS) of 0 or 1
* Histologically confirmed resectable Stage III melanoma according to AJCC-8 and no history of in-transit metastases within the last 6 months
* Fit and planned for CLND
* Measurable disease according to RECIST v1.1
* Availability of a representative tumor specimen
* Adequate hematologic and end-organ function
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative HIV test, negative hepatitis B surface antibody (HBsAb), and negative total hepatitis B core antibody (HBcAb) test, and negative hepatitis C virus (HCV) at screening. Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/μL, and have an undetectable viral load.

Exclusion Criteria for Cohort 1:

* Mucosal, uveal and acral lentiginous melanoma
* Distantly metastasized melanoma
* History of in-transit metastases within the last 6 months
* Prior radiotherapy
* Prior immunotherapy, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, and other systemic therapy for melanoma
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Known immunodeficiency or conditions requiring treatment with systemic immunosuppressive medication, or anticipation of need for systemic immunosuppressant medication during study treatment
* Active or history of autoimmune disease or immune deficiency

Inclusion Criteria for Cohort 2:

* ECOG PS of 0 or 1
* Life expectancy >= 3 months, as determined by the investigator
* Histologically confirmed Stage IV (metastatic) cutaneous melanoma according to AJCC-8
* Disease progression during or following at least one but no more than two lines of treatment for metastatic disease
* Measurable disease according to RECIST v1.1
* Availability of a representative tumor specimen
* Adequate hematologic and end-organ function
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative HIV test, negative hepatitis B surface antibody (HBsAb), and negative total hepatitis B core antibody (HBcAb) test, and negative hepatitis C virus (HCV) at screening. Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/μL, and have an undetectable viral load.

Exclusion Criteria for Cohort 2:

* Mucosal and uveal melanoma
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Known immunodeficiency or conditions requiring treatment with systemic immunosuppressive medication, or anticipation of need for systemic immunosuppressant medication during study treatment
* Active or history of autoimmune disease or immune deficiency
* Symptomatic, untreated, or progressing CNS metastases
* Active or history of carcinomatous meningitis/leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (4):
  - City of Hope, Duarte, California
  - The Angeles Clinic and Research Institute - W LA Office, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - MD Anderson Cancer Center, Houston, Texas
- Melanoma Institute Australia, North Sydney, New South Wales, Australia
- France (4):
  - Hopital de la Timone, Marseille
  - APHP - Hospital Saint Louis, Paris
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (4):
  - Azienda Ospedaliera Universitaria Senese, Siena, Abruzzo
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Ospedale S.Maria della Misericordia, Perugia, Umbria
- Hospital Universitario Vall d Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here ( https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Long GV, Nair N, Marbach D, Scolyer RA, Wilson S, Cotting D, Staedler N, Amaria RN, Ascierto PA, Tarhini AA, Robert C, Hamid O, Gaudy-Marqueste C, Lebbe C, Munoz-Couselo E, Menzies AM, Pages C, Curigliano G, Mandala M, Jessop N, Bader U, Perdicchio M, Teichgraber V, Muecke M, Markert C, Blank C. Neoadjuvant PD-1 and LAG-3-targeting bispecific antibody and other immune checkpoint inhibitor combinations in resectable melanoma: the randomized phase 1b/2 Morpheus-Melanoma trial. Nat Med. 2025 Nov;31(11):3700-3712. doi: 10.1038/s41591-025-03967-2. Epub 2025 Sep 24. PMID 40993242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 14 investigative sites in 5 countries: the United States, Italy, France, Spain, and Australia.
  The study is considered "Completed" because all the pre-planned study activities and analyses have been performed.
Pre-assignment Details: A total of 110 participants with resectable Stage III melanoma and Stage IV melanoma took part in Cohort 1 and Cohort 2, respectively. A total of 6 treatment arms were planned in Cohort 1 and 102 participants were enrolled in only 4 arms. The study was closed before the Cohort 1 arms tobemstomig 600 milligrams (mg), and tobemstomig 600 mg + tiragolumab were opened. 8 participants were enrolled in 1 arm in Cohort 2.
Groups:
- Cohort 1: Nivolumab + Ipilimumab (Control): Participants received nivolumab 3 milligrams/kilograms (mg/kg) intravenously (IV) and ipilimumab 1 mg/kg IV on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first. Post-surgery at the discretion of the investigator, participants started either adjuvant therapy or an observation phase from Week 13.
- Cohort 1: Tobemstomig 2100 mg: Participants received a fixed dose of tobemstomig 2100 mg IV on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first. Post-surgery at the discretion of the investigator, participants started either adjuvant therapy or an observation phase from Week 13.
- Cohort 1: Atezolizumab + Tiragolumab: Participants received atezolizumab 1200 mg IV and tiragolumab 600 mg IV on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first. Post-surgery at the discretion of the investigator, participants started either adjuvant therapy or an observation phase from Week 13.
- Cohort 1: Tobemstomig + Tiragolumab: Participants received tobemstomig 2100 mg IV and tiragolumab 600 mg IV on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first. Post-surgery at the discretion of the investigator, participants started either adjuvant therapy or an observation phase from Week 13.
- Cohort 2: Tobemstomig + Tiragolumab: Participants received tobemstomig 2100 mg IV and tiragolumab 600 mg IV on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
Period: Overall Study
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab | Cohort 2: Tobemstomig + Tiragolumab
Started | 22 | 40 | 20 | 20 | 8
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 22 | 40 | 20 | 20 | 8
Not completed — Study Terminated by Sponsor | 21 | 38 | 17 | 18 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Death | 1 | 1 | 2 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were enrolled in the study.
Groups:
- Cohort 1: Nivolumab + Ipilimumab (Control): Participants received nivolumab 3 mg/kg IV and ipilimumab 1 mg/kg IV on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first. Post-surgery at the discretion of the investigator, participants started either adjuvant therapy or an observation phase from Week 13.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab | Cohort 2: Tobemstomig + Tiragolumab | Total
Number analyzed (Participants) | 22 | 40 | 20 | 20 | 8 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.05 (16.03) | 64.10 (10.97) | 58.90 (14.10) | 59.15 (10.69) | 52.63 (14.22) | 59.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 8 | 6 | 3 | 37
  Male | 11 | 31 | 12 | 14 | 5 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 13 | 29 | 10 | 16 | 8 | 76
  Unknown or Not Reported | 8 | 11 | 10 | 4 | 0 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 15 | 35 | 14 | 14 | 8 | 86
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 6 | 4 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response Rate (pRR) for Cohort 1 as Determined by Independent Pathologic Review
Description: pRR was defined as the percentage of participants with pathologic complete response (pCR), pathologic near complete response (pnCR), and pathologic partial response (pPR) as determined by an independent pathologic review. pCR was defined as a complete absence of viable tumor cells, pnCR as > 0 to ≤ 10% of viable tumor cells, and pPR was defined as > 10 to ≤ 50% of viable tumor cells in the dissected lymph node. Participants with missing or no pathologic response assessment, including participants who did not proceed to complete lymph node dissection (CLND), were classified as non-responders. pRR was calculated for each arm along with 95% confidence intervals (CIs) using Clopper-Pearson method. The difference in pRR between the experimental arms and the control arm was calculated, along with 95% CIs using the Wald method with continuity correction.
Time Frame: Time of surgery (scheduled at Week 7)
Population: Efficacy-evaluable population included all participants in Cohort 1 who received at least one dose of each drug for their assigned treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
percentage of participants | 77.3 [54.63 to 92.18] | 80.0 [64.35 to 90.95] | 45.0 [23.06 to 68.47] | 60.0 [36.05 to 80.88]
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig 2100 mg; Test type: Superiority; Difference in pRR = 2.73, 95% CI 2-sided [-22.25 to 27.70]
Statistical Analysis 2: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Atezolizumab + Tiragolumab; Test type: Superiority; Difference in pRR = -32.27, 95% CI 2-sided [-65.01 to 0.46]
Statistical Analysis 3: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig + Tiragolumab; Test type: Superiority; Difference in pRR = -17.27, 95% CI 2-sided [-49.75 to 15.21]

2. Primary Outcome: Objective Response Rate (ORR) for Cohort 2 as Determined by the Investigator
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in the short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Participants with missing or no response assessments were classified as non-responders. ORR was calculated for each arm, along with 95% CIs using Clopper-Pearson method.
Time Frame: From randomization up to approximately 3.6 months
Population: Efficacy-evaluable population included all participants in Cohort 2 who received at least one dose of each drug for their assigned treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 8
percentage of participants | 0 [0 to 36.94]

3. Secondary Outcome: pRR for Cohort 1 as Determined by Local Pathologic Assessment
Description: pRR was defined as the percentage of participants with pCR, pnCR, and pPR as determined by a local pathologic review. pCR was defined as a complete absence of viable tumor cells, pnCR as > 0 to ≤ 10% of viable tumor cells, and pPR was defined as > 10 to ≤ 50% of viable tumor cells in the dissected lymph node. Participants with missing or no pathologic response assessment, including participants who did not proceed to CLND, were classified as non-responders. pRR was calculated for each arm along with 95% CIs using Clopper-Pearson method. The difference in pRR between the experimental arms and the control arm was calculated, along with 95% CIs using the Wald method with continuity correction.
Time Frame: Time of surgery ( scheduled at Week 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
percentage of participants | 81.8 [59.72 to 94.81] | 75.0 [58.80 to 87.31] | 50.0 [27.20 to 72.80] | 60.0 [36.05 to 80.88]
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig 2100 mg; Test type: Superiority; Difference in pRR = -6.82, 95% CI 2-sided [-31.31 to 17.68]
Statistical Analysis 2: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Atezolizumab + Tiragolumab; Test type: Superiority; Difference in pRR = -31.82, 95% CI 2-sided [-63.79 to 0.16]
Statistical Analysis 3: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig + Tiragolumab; Test type: Superiority; Difference in pRR = -21.82, 95% CI 2-sided [-53.44 to 9.80]

4. Secondary Outcome: Event-free Survival (EFS) for Cohort 1
Description: EFS was defined as the time from randomization to any of the following events (whichever occurs first): documented disease progression (PD) that precludes surgery, as assessed by investigator per RECIST v1.1, local, regional, or distant disease recurrence, or death from any cause. PD = as at least a 20% increase in smallest sum of diameter (SOD) of target lesions, taking as reference the smallest SOD on study (including baseline). Local recurrence was defined as tumor regrowth within 2 cm of the primary lesion's tumor bed; regional recurrence as any nodal or non-nodal tumor lesions that are > 2 cm from the primary lesion but not beyond the regional nodal basin; distant recurrence as any non-local/non-regional recurrence. Participants without disease recurrence, progression, or death at the time of analysis were censored at the time of the last tumor assessment. Kaplan-Meier method was used to estimate the median for EFS, and 95% CIs was constructed using Brookmeyer and Crowley method.
Time Frame: From randomization to disease progression, disease recurrence or death or last tumor assessment (up to 22.51 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
months | 19.55 [19.55 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | NA [14.09 to NA] — The median and upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 22.51 [6.08 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | NA [6.51 to NA] — The median and upper limit of the 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig 2100 mg; Test type: Superiority; Hazard Ratio (HR) = 2.09, 95% CI 2-sided [0.42 to 10.42]
Statistical Analysis 2: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Atezolizumab + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 3.95, 95% CI 2-sided [0.79 to 19.70]
Statistical Analysis 3: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 6.27, 95% CI 2-sided [0.73 to 53.70]

5. Secondary Outcome: Relapse-free Survival (RFS) for Cohort 1
Description: RFS was defined as the time from surgery to the first documented recurrence of disease or death from any cause. Recurrent disease includes local, regional, or distant recurrence: local recurrence was defined as tumor regrowth within 2 cm of the primary lesion's tumor bed; regional recurrence as any nodal or non-nodal tumor lesions that are more than 2 cm from the primary lesion but are not beyond the regional nodal basin; distant recurrence as any non-local/non-regional recurrence. Participants without disease recurrence or death at the time of analysis were censored at the last tumor assessment. Kaplan-Meier method was used to estimate the median for RFS, and 95% CIs were constructed using the Brookmeyer and Crowley method.
Time Frame: From surgery (scheduled at Week 7) to first documented disease recurrence or death or last tumor assessment (up to 20.9 months)
Population: Adjuvant evaluable population included participants in Cohort 1 who had completed surgery (CLND).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 38 | 18 | 19
months | 17.91 [17.91 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 17.08 [11.79 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 20.90 [4.40 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig 2100 mg; Test type: Superiority; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.25 to 7.75]
Statistical Analysis 2: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Atezolizumab + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 2.09, 95% CI 2-sided [0.35 to 12.62]
Statistical Analysis 3: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 2.39, 95% CI 2-sided [0.22 to 26.32]

6. Secondary Outcome: Overall Survival (OS) for Cohort 1
Description: OS was defined as the time from randomization to death from any cause. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. Kaplan-Meier method was used to estimate the median for OS, 95% CIs were constructed using the Brookmeyer and Crowley method.
Time Frame: From randomization to death from any cause or last known to be alive (Up to 25 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
months | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig 2100 mg; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.05 to 12.39]
Statistical Analysis 2: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Atezolizumab + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 2.59, 95% CI 2-sided [0.23 to 28.65]
Statistical Analysis 3: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.07 to 18.58]

7. Secondary Outcome: ORR for Cohort 1
Description: ORR was defined as the percentage of participants with a CR or PR, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Participants with missing or no response assessments were classified as non-responders. ORR was calculated for each arm, along with 95% CIs using the Clopper-Pearson method. The difference in ORR between the experimental arms and the control arm was calculated, along with 95% CIs using the Wald method with continuity correction.
Time Frame: Prior to surgery (up to Week 6)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
percentage of participants | 59.1 [36.35 to 79.29] | 37.5 [22.73 to 54.20] | 35.0 [15.39 to 59.22] | 60.0 [36.05 to 80.88]
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig 2100 mg; Test type: Superiority; Difference in ORR = -21.59, 95% CI 2-sided [-50.55 to 7.37]
Statistical Analysis 2: Comparison: Cohort 1: Atezolizumab + Tiragolumab; Test type: Superiority; Difference in ORR = -24.09, 95% CI 2-sided [-58.17 to 9.99]
Statistical Analysis 3: Comparison: Cohort 1: Nivolumab + Ipilimumab (Control) vs Cohort 1: Tobemstomig + Tiragolumab; Test type: Superiority; Difference in ORR = 0.91, 95% CI 2-sided [-33.58 to 35.40]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Severity of AEs Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0) for Cohort 1
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. Severity was determined per NCI CTCAE v5.0 Grade 1: Mild; asymptomatic or mild symptoms; clinical/diagnostic observations only; or intervention not indicated; Grade 2:Moderate; minimal, local/non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living (ADL); Grade 3: Severe or medically significant, but not immediately life-threatening: hospitalization or prolongation of hospitalization indicated; disabling or limiting self-care ADL; Grade 4: Life-threatening consequences or urgent intervention indicated; Grade 5: Death related to AE. Multiple occurrences of AEs in the same category at the worst (highest) NCIC-CTCAE grade for an individual are counted only once.
Time Frame: From initiation of study treatment up to 135 days (Serious AEs and AESI) or 30 days (all other AEs) after the final dose of study treatment or until initiation of new systemic anti-cancer therapy (Up to 5.6 months)
Population: Safety-evaluable population included all randomized participants in Cohort 1 who received any amount of study treatment. All AEs were reported until 30 days after final dose or until initiation of new systemic anti-cancer therapy (whichever occurs first). Serious AEs and AEs of special interest (AESIs) and treatment-related non-serious AEs that lead to surgery delay were reported until 135 days after final dose or until initiation of new systemic anti-cancer therapy (whichever occurs first).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
Participants
  AE, Any Grade | 19 | 36 | 19 | 18
  Worst Grade, Grade 1 AE | 4 | 13 | 9 | 4
  Worst Grade, Grade 2 AE | 9 | 15 | 9 | 8
  Worst Grade, Grade 3 AE | 4 | 5 | 1 | 6
  Worst Grade, Grade 4 AE | 2 | 3 | 0 | 0
  Worst Grade, Grade 5 AE | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Immune-related AEs Grade ≥ 3 for Cohort 1
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. Participants with immune-related adverse events Grade ≥ 3 were reported.
Time Frame: From initiation of study treatment up to 135 days after the final dose of study treatment (Up to 5.6 months)
Population: Safety-evaluable population included all randomized participants in Cohort 1 who received any amount of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
Participants | 5 | 1 | 0 | 3

10. Secondary Outcome: Rate of Delayed Surgery Due to Treatment-related AEs
Description: Rate of delayed surgery due to treatment related AEs was defined as the percentage of participants for whom surgery was delayed due to treatment-related AEs for more than 2 weeks. An AE was any untoward medical occurrence in a clinical investigation participants administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of the investigational product, whether considered related to the investigational product.
Time Frame: Time of surgery (scheduled at Week 7) up to 40.1 weeks
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 40 | 20 | 20
percentage of participants | 13.6 | 2.5 | 0 | 5.0

11. Secondary Outcome: Duration of Surgery Delay Due to Treatment-related AEs
Description: Duration of surgery delay due to treatment related AEs was calculated on the participants for whom surgery was delayed due to treatment-related AEs for more than 2 weeks. An AE was any untoward medical occurrence in a clinical investigation participants administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with the use of the investigational product, whether considered related to the investigational product.
Time Frame: Time of surgery (scheduled at Week 7) up to 40.1 weeks
Population: Safety-evaluable population included all randomized participants in Cohort 1 who received any amount of the study treatment. Participants with a surgery delay of more than 2 weeks due to treatment-related AE were analyzed.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 3 | 1 | 0 | 1
weeks | 17.0 (14.8) | 5.1 (NA) — The Standard Deviation (SD) was not estimable due to insufficient number of participants with events. |  | 3.0 (NA) — The SD was not estimable due to insufficient number of participants with events.

12. Secondary Outcome: Surgical Complication Rates for Cohort 1
Description: Surgical complications were scored according to the Clavien-Dindo surgical classification. Complication rates for every grade were reported and scored for participants who underwent CLND. The Surgical complications according to Clavien-Dindo can be classified into the following grades: Grade I: Any complication that does not need pharmacological treatment or surgical, endoscopic, and radiological interventions. Grade II: Complications that require pharmacological treatment with drugs or blood transfusions and total parenteral nutrition. Grade III: Complications that require surgical, endoscopic, or radiological intervention with (Grade IIIb) or without (Grade IIIa) general anesthesia. Grade IV: Life-threatening complications requiring intensive care unit (ICU) management, which may be single organ (Grade IVa) or multiorgan (Grade IVb) dysfunction. Grade V: Complications that might cause the death of a participant. Values have been rounded off to 2 decimal digits.
Time Frame: At treatment discontinuation visit (Week 13) and Surgery Follow-Up (6 months after surgery)
Population: Safety-evaluable population included all randomized participants in Cohort 1 who received any amount of the study treatment. Overall number analyzed is the number of participants who underwent surgery. Number analyzed is the number of participants with surgical complication.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 22 | 38 | 18 | 19
percentage of participants
  Treatment Discontinuation Visit: Grade 0 | 0 | 0 | 5.55 | 5.26
  Treatment Discontinuation Visit: Grade I | 18.18 | 5.26 | 22.22 | 0
  Treatment Discontinuation Visit: Grade II | 13.63 | 18.42 | 16.66 | 10.52
  Treatment Discontinuation Visit: Grade IIIa | 0 | 7.89 | 0 | 5.26
  Treatment Discontinuation Visit: Grade IIIb | 0 | 2.63 | 0 | 10.52
  Treatment Discontinuation Visit: Grade IVa | 0 | 2.63 | 0 | 0
  Long-term Follow-up Month 6: Grade 0: number analyzed (Participants) | 22 | 37 | 17 | 17
  Long-term Follow-up Month 6: Grade 0 | 0 | 0 | 5.88 | 0
  Long-term Follow-up Month 6: Grade I: number analyzed (Participants) | 22 | 37 | 17 | 17
  Long-term Follow-up Month 6: Grade I | 13.63 | 8.11 | 17.64 | 0
  Long-term Follow-up Month 6: Grade II: number analyzed (Participants) | 22 | 37 | 17 | 17
  Long-term Follow-up Month 6: Grade II | 4.54 | 10.81 | 5.88 | 0
  Long-term Follow-up Month 6: Grade IIIa: number analyzed (Participants) | 22 | 37 | 17 | 17
  Long-term Follow-up Month 6: Grade IIIa | 0 | 13.51 | 5.88 | 0
  Long-term Follow-up Month 6: Grade IIIb: number analyzed (Participants) | 22 | 37 | 17 | 17
  Long-term Follow-up Month 6: Grade IIIb | 0 | 0 | 0 | 11.76
  Long-term Follow-up Month 6: Grade IVa: number analyzed (Participants) | 22 | 37 | 17 | 17
  Long-term Follow-up Month 6: Grade IVa | 0 | 2.7 | 0 | 0

13. Secondary Outcome: Progression-Free Survival (PFS) for Cohort 2
Description: PFS after randomization/enrollment was defined as the time from randomization/enrollment to the first occurrence of disease progression or death from any cause (whichever occurred first), as determined by the investigator according to RECIST v1.1. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on the study (including baseline) and/or unequivocal progression of a non-target lesion and/or any new lesion. Participants without documented disease progression or death at the time of analysis were censored at the day of the last tumor assessment. Kaplan-Meier method was used to estimate the median for PFS, with 95% CIs constructed by using the Brookmeyer and Crowley method.
Time Frame: From randomization/enrollment to first documented disease progression or death or last tumor assessment (up to 3.6 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 8
months | 2.07 [1.68 to 2.37]

14. Secondary Outcome: OS for Cohort 2
Description: OS was defined as the time from randomization to death from any cause. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. Kaplan-Meier method was used to estimate the median for OS, with 95% CIs constructed by using the Brookmeyer and Crowley method.
Time Frame: From randomization/enrollment to death from any cause or last known to be alive (Up to 24.2 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 8
months | 8.94 [4.17 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

15. Secondary Outcome: OS Rates at Specific Timepoints for Cohort 2
Description: OS was defined as the time from randomization to death from any cause. OS rate is percentage of participants who were event free for OS. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. OS rate at specific time points were estimated using the Kaplan-Meier method, with 95% CIs calculated based on Greenwood's estimate for the variance.
Time Frame: Months 3, 6 and 12
Population: Efficacy-evaluable population included all participants in Cohort 2 who received at least one dose of each drug for their assigned treatment regimen. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an OS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 8
percentage of participants
  3 months: number analyzed (Participants) | 7
  3 months | 100.0 [100.0 to 100.0]
  6 months: number analyzed (Participants) | 4
  6 months | 71.43 [37.96 to 100.0]
  12 months: number analyzed (Participants) | 2
  12 months | 47.62 [3.47 to 91.77]

16. Secondary Outcome: Duration of Response (DOR) for Cohort 2
Description: DOR was defined as the time from the first occurrence of a documented objective response (OR) to disease progression or death from any cause (whichever occurred first), as determined by the investigator according to RECIST v1.1. OR was defined as a CR or PR on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR = disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR = at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on the study (including baseline). Participants without PD or death at time of analysis were censored at time of last tumor assessment. Kaplan-Meier method was used to estimate median for DOR, with 95% CIs constructed using Brookmeyer & Crowley method.
Time Frame: Time from the first occurrence of a documented OR to disease progression or death from any cause (up to 3.6 months)
Population: Efficacy-evaluable population included all participants in Cohort 2 who received at least one dose of each drug for their assigned treatment regimen.
  DOR was only evaluated in participants who achieved an OR (CR or PR).
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Disease Control Rate (DCR) for Cohort 2
Description: DCR was defined as the percentage of participants with stable disease for ≥ 12 weeks or a CR or PR, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Stable disease was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on the study (including baseline). DCR was calculated for each treatment arm, with 95% CIs estimated through use of Clopper-Pearson's exact method.
Time Frame: From randomization up to 3.6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 8
percentage of participants | 0 [0.00 to 36.94]

18. Secondary Outcome: Number of Participants With AEs and Severity of AEs Determined According to NCI CTCAE v5.0 for Cohort 2
Description: An AE=any untoward medical occurrence in clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. AE can therefore be any unfavorable & unintended sign, symptom/disease temporally associated with using an investigational product, whether or not considered related to the investigational product. Severity was determined per NCI CTCAE v5.0 Grade 1: Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; or intervention not indicated; Grade 2: Moderate; minimal, local/non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living (ADL); Grade 3: Severe/medically significant, but not immediately life-threatening: hospitalization/prolongation of hospitalization indicated; disabling/limiting self-care ADL; Grade 4: Life-threatening consequences/urgent intervention indicated; Grade 5: Death related to AE. Multiple occurrences of AEs in 1 individual are counted once at highest grade.
Time Frame: From initiation of study treatment up to 135 days (Serious AEs and AESI) or 30 days (all other AEs) after the final dose of study treatment or until initiation of new systemic anti-cancer therapy (Up to 10 months)
Population: Safety-evaluable population included all randomized participants in Cohort 2 who received any amount of the study treatment. All AEs were reported until 30 days after the final dose or until initiation of new systemic anti-cancer therapy (whichever occurs first). Serious AEs and AESIs were reported until 135 days after the final dose or until initiation of new systemic anti-cancer therapy (whichever occurs first).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Tobemstomig + Tiragolumab
Number analyzed (Participants) | 8
Participants
  AE, Any Grade | 7
  Worst Grade, Grade 1 AE | 0
  Worst Grade, Grade 2 AE | 6
  Worst Grade, Grade 3 AE | 1
  Worst Grade, Grade 4 AE | 0
  Worst Grade, Grade 5 AE | 0

ADVERSE EVENTS:
Time Frame: From initiation of study treatment up to 135 days (Serious AEs and AESI) or 30 days (all other AEs) after the final dose of study treatment or until initiation of new systemic anti-cancer therapy (Up to 5.6 months for Cohort 1 and 10 months for Cohort 2); All-cause Mortality: Randomization up to the end of long-term follow-up (Up to approximately 25 months for Cohort 1 and 24.2 months for Cohort 2)
Description: Safety evaluable population included all randomized participants who received at least one dose of the study drug.
Arm/Group | Cohort 1: Nivolumab + Ipilimumab (Control) | Cohort 1: Tobemstomig 2100 mg | Cohort 1: Atezolizumab + Tiragolumab | Cohort 1: Tobemstomig + Tiragolumab | Cohort 2: Tobemstomig + Tiragolumab
All-Cause Mortality (participants affected / at risk) | 1/22 | 1/40 | 2/20 | 1/20 | 5/8
Serious Adverse Events (participants affected / at risk) | 4/22 | 9/40 | 3/20 | 6/20 | 1/8
Other Adverse Events (participants affected / at risk) | 18/22 | 34/40 | 18/20 | 18/20 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Nivolumab + Ipilimumab (Control) (N=22) | Cohort 1: Tobemstomig 2100 mg (N=40) | Cohort 1: Atezolizumab + Tiragolumab (N=20) | Cohort 1: Tobemstomig + Tiragolumab (N=20) | Cohort 2: Tobemstomig + Tiragolumab (N=8)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphatic fistula (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Nivolumab + Ipilimumab (Control) (N=22) | Cohort 1: Tobemstomig 2100 mg (N=40) | Cohort 1: Atezolizumab + Tiragolumab (N=20) | Cohort 1: Tobemstomig + Tiragolumab (N=20) | Cohort 2: Tobemstomig + Tiragolumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 7 (7) | 3 (3) | 6 (6) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (5) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (7) | 15 (15) | 3 (4) | 6 (6) | 4 (4)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (4)
Xerosis (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Contrast media allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 6 (8) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 8 (8) | 4 (4) | 3 (3) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (6) | 2 (2) | 5 (5) | 2 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (8) | 1 (1) | 3 (3) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsorâ€™s intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05116202/Prot_SAP_000.pdf